CLINICAL TRIAL: NCT05341180
Title: Efficacy of Polyethylene Glycol vs Lactulose With Isabgol in Acute Fissure-in-Ano: A Randomized Control Trial (PEGASIS Trial)
Brief Title: Efficacy of Polyethylene Glycol vs Lactulose With Isabgol in Acute Fissure-in-Ano: PEGASIS Trial
Acronym: PEGASIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Prakash Kumar Sasmal, Additional Professor, Department of General Surgery, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC/AIIMS BBSR/PG Thesis/
Record Dates: First submitted 2022-04-10; First posted 2022-04-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Anal Fissure; Constipation
Keywords: Acute fissure in ano; Constipation; Lactulose; Isabgol; Polyethylene Glycol
MeSH Terms: conditions — Fissure in Ano; Constipation | interventions — Polyethylene Glycols; Lactulose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1(Polyethylene Glycol) (Active Comparator): Polyethylene glycol syrup will be used at a dose of 15-30 ml per day for 2 weeks maximum.
  Interventions: Drug: Polyethylene Glycol
- Study group 2 (Isabgol and Lactulose) (Active Comparator): Isabgol 2 teaspoons in 200ml of warm water to consume immediately after soaking before bedtime and syrup Lactulose 30 ml at bedtime for 2 weeks.
  Interventions: Drug: Isabgol + Lactulose

INTERVENTIONS:
Drug: Polyethylene Glycol — Patients will be advised Anobliss (lidocaine with nifedipine) ointment for local application in the anal canal for one month for relief of pain and anal sphincter spasm. Polyethylene glycol syrup at a dose of 15-30 ml will be used for 2 weeks for relief of acute constipation. Patients will be assessed at 1 week and 1 month and evaluated for primary and secondary outcomes.
  Other Names: Freego PEG oral solution from Alembic Pharmaceuticals Ltd.
  Arms: Study group 1(Polyethylene Glycol)
Drug: Isabgol + Lactulose — Patients will be advised Anobliss (lidocaine with nifedipine) ointment for local application in the anal canal for one month for relief of pain and anal sphincter spasm. Isabgol husk at a dose of 2 teaspoons in 200 ml of warm water before bedtime and 30 ml of syrup lactulose at bedtime will be used for 2 weeks for relief of acute constipation. Patients will be assessed at 1 week and 1 month and evaluated for primary and secondary outcomes.
  Other Names: Duphalac oral solution from Abbott
  Arms: Study group 2 (Isabgol and Lactulose)

SUMMARY:
The existing literature stresses the better efficacy of polyethylene glycol (PEG) over other stool softeners like lactulose or isabgol to improve functional constipation.

But there is no consensus regarding the efficacy of PEG alone vs lactulose combined with isabgol used as stool softeners, frequently used for relieving acute constipation in an acute fissure in ano. Hence a good quality randomised study to compare both efficacies is the need of the hour.

DETAILED DESCRIPTION:
Acute fissure in ano is a very common, painful and distressing benign anorectal disorder. It is a linear tear in the anoderm of the distal anal canal most commonly on the posterior midline. They usually result from trauma caused by the passage of hard stool and less commonly from diarrhoea also. The most common presenting symptom is anal pain, bleeding and secondary constipation. Most of the cases are managed conservatively by increasing oral fluid intake, high fibre diet, sitz bath, stool softeners and topical application of sphincter muscle relaxants.

Constipation is one of the most common causes of anal fissure. Patients present to the outpatient department due to acute anal pain resulting from increased internal anal sphincter tone with spasms and hard stool rubbing over the crack. Constipation and pain due to anal fissure are initially managed with lifestyle and dietary modifications like consuming adequate fluids, increased fibre diet and sitz bath.

One of the fibre supplements is isabgol husk, a soluble fibre with enormous water-absorbing properties. Its added benefits include properties like non-irritant to the large bowel, non-fermenting, and dichotomous stool normalising agents, making it one of the most preferred bulk-forming agents. Low cost and over the counter availability are other benefits. Lactulose is also the most commonly prescribed laxative used in acute anal fissures to relieve constipation. Polyethylene glycol is a common osmotic laxative used for the relief of constipation in the treatment of anal fissures.

There are multiple studies that say polyethylene glycol has better efficacy in terms of frequency of stools, and form of stools compared to lactulose or isabgol husk alone. However, there are no studies conducted to compare the efficacy of polyethylene glycol vs combined use of isabgol husk and lactulose in relief of constipation in an acute fissure in ano. However, studies prove that laxatives may reduce/delay the absorption of certain medications, hence medications are advised to be taken 1 hour before or 2-3 hours after taking laxatives.

Patients in both arms will be advised to use local lidocaine with nifedipine cream (Anobliss cream from Samarth Life Sciences Pvt. Ltd., India). One arm will be given polyethylene glycol syrup for 2 weeks maximum and in the other arm, isabgol husk plus lactulose will be given for 2 weeks. Patients will be assessed at the end of a week, and 1 month and evaluated for primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with acute fissure in ano between the age group of 18 to 75 years.

Exclusion Criteria:

* Pregnancy / lactation

  * Patients not giving consent
  * Patients not able to understand the nature of the study
  * Diabetes mellitus and chronic kidney disease
  * Known intolerance to PEG/Lactulose or Isabgol
  * Prior enrolment in other study.
  * Patient undergoing surgery for Fissure in Ano

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Time taken for the resolution of acute pain following fissure in ano. | 30 days
  Pain will be measured by improvement in visual analog scale (VAS) pain score. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 10).

SECONDARY OUTCOMES:
Improvement in constipation will be assessed by a change in the Bristol stool form scale. | 1 week, 1 month
  Acute constipation is the cause and result of acute fissure-in-ano. Stool softeners help in alleviating the pain by improving the stool forms assessed by Bristol stool scale. Type 1-2 indicates constipation that exacerbates the pain in an acute fissure in ano. Type 3-4 are ideal stools and easier to pass and Type 5-7 are soft to liquid stools that will be much helpful in alleviating the pain in an acute fissure in ano.
Adverse effects any of PEG or lactulose with isabgol. | 1 month
  Long term use of PEG or lactulose can result in electrolyte imbalance, diarrhoea, or stomach cramps. Incidence of adverse effects if any will be recorded and reported.
Patient compliance with the medications | 1 month
  The compliance with the drugs will be recorded at the end of one month through personal interviews based on TSQM version 1.4 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Kumar Sasmal, MBBS, MS, Principal Investigator — Department of General Surgery, All India Institute of Medical Sciences, Bhubaneswar, Odisha, INDIA
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee-Robichaud H, Thomas K, Morgan J, Nelson RL. Lactulose versus Polyethylene Glycol for Chronic Constipation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007570. doi: 10.1002/14651858.CD007570.pub2. PMID 20614462
- [Background] Wang HJ, Liang XM, Yu ZL, Zhou LY, Lin SR, Geraint M. A Randomised, Controlled Comparison of Low-Dose Polyethylene Glycol 3350 plus Electrolytes with Ispaghula Husk in the Treatment of Adults with Chronic Functional Constipation. Clin Drug Investig. 2004;24(10):569-76. doi: 10.2165/00044011-200424100-00002. PMID 17523718
- [Background] Tomatsu S, Dieter T, Schwartz IV, Sarmient P, Giugliani R, Barrera LA, Guelbert N, Kremer R, Repetto GM, Gutierrez MA, Nishioka T, Serrato OP, Montano AM, Yamaguchi S, Noguchi A. Identification of a common mutation in mucopolysaccharidosis IVA: correlation among genotype, phenotype, and keratan sulfate. J Hum Genet. 2004;49(9):490-494. doi: 10.1007/s10038-004-0178-8. Epub 2004 Aug 11. PMID 15309681
- [Background] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789
- [Background] Belsey JD, Geraint M, Dixon TA. Systematic review and meta analysis: polyethylene glycol in adults with non-organic constipation. Int J Clin Pract. 2010 Jun;64(7):944-55. doi: 10.1111/j.1742-1241.2010.02397.x. PMID 20584228

DOCUMENTS (1):
  • Study Protocol (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05341180/Prot_001.pdf